CLINICAL TRIAL: NCT07099885
Title: Simple Urine Composition-based Personalized Algorithm for Effective Congestion Relief in Decompensated Heart Failure
Acronym: SAFER-DHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jan Biegus, MD, PhD, Professor, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 226/2025
Record Dates: First submitted 2025-07-15; First posted 2025-08-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Heart Failure (AHF); Congestion, Venous
Keywords: decongestion; diuretics; algorithm; acute heart failure
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithm based decongestion (Experimental): The patient will receive first dose of intravenous loop diuretic determined per the attending physician. Two hours after diuretic administration, a urine sample will be collected to measure sodium and creatinine concentrations. Using these values, the 6-hour urine output will be estimated with the aid of the machine learning, urine output prediction tool. This estimated diuresis will guide the diuretic therapy plan for the first 24 hours using the adaptative furosemide dosing.
  On the second day, the procedure will be repeated.
  Interventions: Diagnostic Test: Algorithhm-based decongestion
- Standard of care (Active Comparator)
  Interventions: Diagnostic Test: Standard of Care (SOC)

INTERVENTIONS:
Diagnostic Test: Standard of Care (SOC) — Diuretic treatment per attending physician.
  Arms: Standard of care
Diagnostic Test: Algorithhm-based decongestion — Patient will receive standarized furosemide dosing based on the result of the algorithm-estimated 6h urine output (profiles of diuretic response).
  Arms: Algorithm based decongestion

SUMMARY:
The aim of this study is to evaluate the effectiveness of loop diuretic adaptative algorithm that is based on machine learning, urine output prediction tool, in decongestion of acute heart failure patients.

A total of 90 patients will be enrolled in the study. Of these, 45 will be assigned to the algorithm-based intervention group, while the remaining 45 will serve as the control group. In the control group, all decisions regarding diuretic therapy will be made solely by the attending physician, without the use of the algorithm.

Patients will receive intravenous furosemide, with the initial dose determined by the attending physician. Two hours after administration of the diuretic, a spot urine sample will be collected to measure sodium and creatinine concentrations. Based on these values, the 6-hour urine output will be estimated using the machine learning, urine output prediction tool (http://diuresis.umw.edu.pl). This estimate will guide the diuretic therapy plan for the first 24 hours of hospitalization. On the second day, the procedure will be repeated using the same methodology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who provide informed consent
* Ability to enroll in the study within the first 24 hours of hospitalization
* Primary reason for hospitalization is acute heart failure with signs of congestion (at least moderate lower extremity edema)
* NT-proBNP > 1500 pg/ml
* Anticipated need for diuretic therapy for at least 48 hours from the time of study enrollment

Exclusion Criteria:

* End-stage kidney disease requiring renal replacement therapy
* Hemodynamic instability requiring inotropic support
* Active infection requiring intravenous antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative diuresis over 48 hours. | 48 hours
  Total urine output during the 48-hour duration of the study.

SECONDARY OUTCOMES:
Cumulative diuresis during first 24h of the study. | 24 hours
  The total urine output during the first 24 hours of the study.
Cumulative diuresis on the second 24h of the study. | 48 hours
  The total urine output during the second 24 hours of the study.
Cummulative natriuresis over 48 hours of the study. | 48 hours
  The total amount of sodium excreted in the urine during the 48-hour duration of the study.
Diuresis calculated per dose of loop diuretic over 48 hours of the study. | 48 hours
  The volume of urine output relative to the total dose of loop diuretic administered during the study period.
Weight change at 24 hours. | 24 hours
  The difference in body weight measured at 24 hours compared to baseline.
Weight change at 48 hours. | 48 hours
  The difference in body weight measured at 48 hours compared to baseline.
Total length of hospitalization. | Up to 60 days
  This refers to the total length of the hospital stay, measured in days, from admission to discharge.
Percentage of patients accurately red-flagged. | 48 hours
  Patients with an estimated 6-hour urine output of less than 900 ml will be red-flagged. This outcome indicates the proportion of patients who were correctly identified (red-flagged) as poor diuretic responders.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Wroclaw Medical University, Wroclaw, Dolnosląskie
  - Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No